CLINICAL TRIAL: NCT03127007
Title: A Phase Ib/II Study to Evaluate Safety and Efficacy of Atezolizumab Combined With Radio-chemotherapy in a Preoperative Setting for Patients With Localized Rectal Cancer
Brief Title: Safety and Efficacy of Atezolizumab Combined to Preoperative Radio-chemotherapy in Localized Rectal Cancer
Acronym: R-IMMUNE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grand Hôpital de Charleroi (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCOGHdC2015_02
Record Dates: First submitted 2017-04-11; First posted 2017-04-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Rectal Neoplasms
Keywords: immunotherapy; anti-PD-L1
MeSH Terms: conditions — Rectal Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Protracted IV 5-FU 225 mg/m2 is given from day 1 to 5 in parallel with radiotherapy 1.8 to 2 Gy from day 1 to 5 during 5 consecutive weeks.
  Atezolizumab is given on day 1 of week 3, 6, 9 and 12 at 1200 mg IV. Rectal surgery is planned during week 15
  Interventions: Drug: Atezolizumab; Drug: 5-FU based radio-chemotherapy
- Arm B (Active Comparator): Protracted IV 5-FU 225 mg/m2 is given from day 1 to 5 in parallel with radiotherapy 1.8 to 2 Gy from day 1 to 5 during 5 consecutive weeks.
  Rectal surgery is planned during week 15
  Interventions: Drug: 5-FU based radio-chemotherapy

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is given on day 1 of week 3, 6, 9 and 12 at 1200 mg IV.
  Other Names: Tecentriq, MPDL3280a
  Arms: Arm A
Drug: 5-FU based radio-chemotherapy — IV protracted 5-FU given at 225mg/m2 over 24h 5 days/week for 5 weeks associated to radiotherapy.

SUMMARY:
The study has a phase Ib and a phase II part. The phase Ib part of the study aims to determine the safety and tolerance of administration at a fixed dosing of 1200 mg / 3 weeks, concomitantly to the standard preoperative radio-chemotherapy.

The phase II part of the study aims to explore efficacy of atezolizumab in combination with the standard preoperative chemo/radiotherapy in stage II and III rectal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization are obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Male or female > 18 years at time of study entry
* Patients with previously untreated localized T3-T4 N0 or T any or N1-2, M0 rectal adenocarcinoma requiring preoperative radiotherapy
* Availability of protocol required screening tumor and blood samples
* ECOG performance status of 0 or 1
* Adequate normal organ and marrow function:

  1. haemoglobin ≥ 9.0 g/dL, absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3), platelet count ≥ 100 x 109/L (>100,000 per mm3).
  2. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
  3. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit
  4. Serum creatinine CL > 30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 6 months after the last dose of atezolizumab / radio-chemotherapy
* Patients who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Patient has locally recurrent or metastatic RC
* Patient has received any systemic therapy (e.g. chemotherapy, targeted therapy, immunotherapy) or radiotherapy for current rectal cancer disease
* Patients not requiring preoperative radio-chemotherapy
* Participation in another clinical study with an investigational product for any other indication until 4 weeks before study participation
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 21 days prior to the first dose of study drug
* Any previous treatment with a PD1 or PD-L1 inhibitor, including atezolizumab
* History of another primary malignancy except for:

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
* Current or prior use of immunosuppressive medication within 28 days before the first dose of atezolizumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to randomization
* Receipt of live attenuated vaccination within 30 days prior first atezolizumab planned administration (i.e. at week 3 after study entry) or within 5 months of receiving atezolizumab or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination (inactivated forms only but not live attenuated forms) should be given during influenza season only (approximately October to March).
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study. Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to atezolizumab or any excipient
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Subjects with uncontrolled seizures.
* Known history of active tuberculosis
* Female subjects who are pregnant, breast-feeding or female patients of reproductive potential who are not employing or willing to employ an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events | 74 weeks
  Evaluation of adverse events use CTCAE v4.0 terminology
Rate of complete pathological response | 15 weeks
  Evaluation by central pathological review of rectal tumor resected after the preoperative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Javier Carrasco, MD, PhD, Principal Investigator — GHdC; Marc Van den Eynde, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (5):
- Belgium (5):
  - GHdC, Charleroi, Hainaut
  - Katholiek universiteit Leuven, Leuven, Vlaams Brabant
  - Institut Jules Bordet, Brussels
  - Hôpital Erasme, Brussels
  - Cliniques universitaires St Luc, Brussels

IPD SHARING:
Plan to Share IPD: No